CLINICAL TRIAL: NCT01042964
Title: An Open-Label, Dose-Escalating Safety and Pharmacokinetic Study of an Acute Intravenous Administration of PR-15, an Inhibitor of Platelet Adhesion, in Six Different Strengths in Healthy Male Volunteers
Brief Title: Safety, Pharmacokinetic and -Dynamic Study of PR-15, an Inhibitor of Platelet Adhesion
Acronym: PR-15/01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AdvanceCor GmbH (Industry)
Collaborators: Procorde GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-15/01; EudraCT 2005-004656-12 (Registry Identifier: EudraCT)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Thrombosis; Acute Coronary Syndrome; Myocardial Infarction; Stroke
Keywords: platelet adhesion and aggregation; acute coronary syndrome; myocardial infarction; stroke; inhibition of platelet adhesion to plaques; collagen-induced platelet aggregation
MeSH Terms: conditions — Thrombosis; Acute Coronary Syndrome; Myocardial Infarction; Stroke | interventions — Revacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: revacept (PR-15) — single intravenous administration of revacept (PR-15), an inhibitor of platelet adhesion, in various strengths (10, 20, 40, 80, 160 mg) in healthy male volunteers.
  Other Names: GPVI-Fc dimer

SUMMARY:
Primary objective:

To evaluate safety and tolerability, adverse events (AEs), vital signs, ECG, bleeding time, evaluation of antibody titer and safety laboratory tests

Secondary objectives:

To evaluate the pharmacokinetics and pharmacodynamics (platelet aggregation)of six ascending single intravenous doses of PR-15 in healthy volunteers

DETAILED DESCRIPTION:
Primary objective:

To evaluate safety and tolerability by using adverse events (AEs), vital signs including blood pressure/pulse rate (BP/PR), electrocardiographic examinations (12 lead ECG), bleeding time, evaluation of antibody titer and safety laboratory tests (biochemistry, hematology, coagulation, urinalysis)

Secondary objectives:

To evaluate the pharmacokinetics and pharmacodynamics (collagen-induced platelet aggregation)of six ascending single intravenous doses of PR-15 in healthy, male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male Caucasians between 18 and 45 years of age.
* Normotensive subjects (systolic BP < 140 mmHg and diastolic BP <90 mmHg;
* Body weight of 70 to 90 kg (BMI 20 - 25.
* Negative results in HIV antibody, HBs antigen (HBsAg) and HCV tests;
* Signed Informed Consent Form.
* Normal coagulation function (aPTT between 24 and 35 seconds, PT between 70 and 130%, INR between 0.85 and 1.15.

Exclusion Criteria:

* Subjects who are taking or have taken any prescription medication within the last 14 days or any non-prescription medication, especially, anti-platelet drugs, within the last seven days prior to the administration of trial medication on Day 1.
* Intake of any investigational drug within three months prior to the administration of study medication on Day 1.
* Concomitant use of any other medication including over-the-counter preparations.
* History of hypersensitivity, contraindication or serious adverse reaction to inhibitors of platelet aggregation or hypersensitivity to related drugs (cross-allergy) or to any of the excipients in the study drug.
* A history or clinical evidence of any cardiac, cardio- or cerebrovascular, hepatic, renal, pulmonary, endocrine, neurological, infectious, gastrointestinal, haematological, oncological or psychiatric disease or emotional problems or any other clinically relevant condition, physical finding, ECG- or laboratory test abnormality, which - in the opinion of the investigator - would pose a significant risk for the subject, invalidate the Informed Consent or limit the ability of the subject to comply with study requirements or interfere otherwise with the conduct of the study.
* Any laboratory value outside the normal laboratory reference range at Screening and before randomization, unless approved by the investigator.
* Subjects known to have experienced elevated liver enzyme values will also be excluded.
* History of alcohol and/or drug abuse (verified by drug screening).
* Blood loss of 450 ml or more during the last three months before Screening.
* Subjects who smoke more than 5 cigarettes per day and/or are unable to abstain from smoking during the entire in-house period.
* Subjects who were previously enrolled in this trial or who have received PR-15 in a previous trial.
* Subjects who have participated in other clinical trials in the last 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03; Primary Completion 2007-01 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
safety and tolerability adverse events (AEs), vital signs (BP/PR), 12 lead ECG, bleeding time, antibody titer and safety laboratory tests | 43 days

SECONDARY OUTCOMES:
pharmacokinetics and pharmacodynamics (agonist-induced platelet aggregation) | 43 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Piechatzek, MD, Principal Investigator — ABX-CRO/Medifacts GmbH
Locations (1):
- ABX-CRO/Medifacts GmbH, Görlitz, Saxony, Germany

REFERENCES:
- [Result] Ungerer M, Rosport K, Bultmann A, Piechatzek R, Uhland K, Schlieper P, Gawaz M, Munch G. Novel antiplatelet drug revacept (Dimeric Glycoprotein VI-Fc) specifically and efficiently inhibited collagen-induced platelet aggregation without affecting general hemostasis in humans. Circulation. 2011 May 3;123(17):1891-9. doi: 10.1161/CIRCULATIONAHA.110.980623. Epub 2011 Apr 18. PMID 21502572